CLINICAL TRIAL: NCT02816450
Title: The Effects of Hydration on Brain, Cognition, Memory & Achievement in Childhood
Brief Title: Water Intervention for Thinking in Kids (WITiKids ) Study
Acronym: WITiKids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Naiman Khan, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 14701
Record Dates: First submitted 2016-06-17; First posted 2016-06-28 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Low Fluid Intake, Chronic
Keywords: Water; Children; Cognition; Hydration
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Drinking

ARMS (2):
- HIGH (Experimental): Increase water intake to 2.5 liters per day for 4 days
  Interventions: Behavioral: Water Intake
- LOW (Experimental): Decrease water intake to 0.5 liter per day for 4 days
  Interventions: Behavioral: Water Intake

INTERVENTIONS:
Behavioral: Water Intake

SUMMARY:
The aim of this study is to determine the influence of changes in water intake on changes in cognitive function among preadolescent children. Further, the proposed work will determine the relationship between urinary markers of hydration process and cognitive function. We hypothesize that an increase in water intake will result in greater cognitive performance. In addition, improvements in hydration demonstrated by lower urine concentration will be correlated with greater cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

1. Parental/guardian consent
2. Normal or corrected-to-normal vision based on the minimal 20/20 standard in order to complete the cognitive task (below 20/20 vision).

Exclusion Criteria:

1. Participants younger than 9 years and older than 10 years at the time of testing age.
2. Prior diagnosis of cognitive or physical disability, including ADHD (severe asthma, epilepsy, chronic kidney disease, and dependence upon a wheelchair/walking aid).
3. Use of anti-psychotic, anti-depressant, anti-anxiety medication, as well as those medications used for ADD/ADHD (use of any anti-psychotic, anti-depressant, anti-anxiety, and ADD/ADHD medications).
4. Participants must have not yet reached, or be in the earliest stages, of puberty, as measured by a modified test of the Tanner Staging System
5. IQ below 85
6. Use of medications that alter urinary excretion and water metabolism
7. Use of internal electronic device, such as a pacemaker

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Flanker Task Accuracy | 2 Hours on the morning of Day 5

SECONDARY OUTCOMES:
Urine Osmolality | 24 hours during final day of fluid intake modulation (Day 4)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Kinesiology and Community Health, Urbana, Illinois, United States

REFERENCES:
- [Derived] Khan NA, Westfall DR, Jones AR, Sinn MA, Bottin JH, Perrier ET, Hillman CH. A 4-d Water Intake Intervention Increases Hydration and Cognitive Flexibility among Preadolescent Children. J Nutr. 2019 Dec 1;149(12):2255-2264. doi: 10.1093/jn/nxz206. PMID 31504690